CLINICAL TRIAL: NCT01462240
Title: Prospective Multicenter Post-market Study of the Zimmer NexGen LPS-Flex Porous Femoral Components
Brief Title: LPS Flex Porous Femoral Components
Status: Withdrawn | Type: Observational
Why Stopped: Suspended pending internal review/direction of the company's focus.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2010-27K
Record Dates: First submitted 2011-10-24; First posted 2011-10-31 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Poly Arthritis; Collagen Disorders; Avascular Necrosis of Femoral Condyle
Keywords: arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Collagen Diseases; Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 - LPS Flex Pororus Femoral Components: Patients suffering from severe knee pain and disability.
  Interventions: Device: LPS Flex Porous Femoral Components

INTERVENTIONS:
Device: LPS Flex Porous Femoral Components — Porous femoral components in total knee arthroplasty

SUMMARY:
This is a prospective multicenter study of the LPS-Flex Porous Femoral Components when used in primary total knee arthroplasty. The purpose of the study is to obtain short-, mid-, and long-term clinical outcomes and implant survivorship data for the NexGen LPS-Flex Porous Femoral components.

DETAILED DESCRIPTION:
Survival and outcome data on the NexGen LPS-Flex Porous Femoral Components will be done by an analysis of standard scoring system, radiographs and adverse event records. Survivorship will be evaluated by monitoring the frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated adverse device effects. Outcomes will be measured by comparing the overall pain and function performances (based on the Knee Society Scoring System), survivorship, subject quality of life and radiographic parameters of study subjects receiving the LPS-Flex Porous Femoral Components.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18-75 years of age, inclusive;
* Patient qualifies for a total knee arthroplasty based on physical exam and medical history including at least one of the following: rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis, collagen disorders, avascular necrosis of the femoral condyle;
* Post-Traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy;
* Moderate valgus, varus, or flexion deformities;
* Patient has undergone a study related informed consent process;
* Patient is willing and able to provide written consent;
* Patient is willing and able to cooperate in the required post-operative therapy;
* Patient is willing and able to complete scheduled follow-up evaluations.

Exclusion Criteria:

* Patient has previous history of infection in the affected joint and/or a local or systemic infection that could affect the prosthetic joint;
* Insufficient bone stock on femoral or tibial surfaces;
* Skeletal immaturity;
* Neuropathic arthropathy;
* Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb;
* Stable, painless arthrodesis in a satisfactory functional position;
* Severe instability secondary to the absence of collateral ligament integrity;
* Patient has rheumatoid arthritis and an ulcer of the skin or a history of recurrent breakdown of the skin because of their risk of postoperative infection is greater;
* Patient has a known sensitivity or allergy to one or more of the implanted materials;
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mental incompetence, unable to understand what clinical trial participation entails, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each investigator will screen from this patient populatin patients suffering from severe knee pain and disability who meet the inclusion/exclusion criteria for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05-20 (Actual); Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Survivorship | 10 Years
  Based on frequency of adverse events, serious adverse events, adverse device effects, serious adverse device effects and unanticipated adverse device effects or removal of the device summarized using a Kaplan-Meier method and presented with rates (as percentages) and confidence intervals.

SECONDARY OUTCOMES:
Pain and Functional Performance | 10 years
  Measured by comparing the overall pain and function performances (based on Knee Society Scoring System), survivorship, subject quality of life and radiographic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, RN, MBA, Study Director — Zimmer Biomet

IPD SHARING:
Plan to Share IPD: No